CLINICAL TRIAL: NCT06514924
Title: Young Turkish Adults Show a Continuing Positive Secular Change of Height But a Worrying Increase of Overweight in Males
Brief Title: Secular Change of Height in Turkish Young Adults
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ozge Bayrak Demirel, Principal Investigator, Istanbul University
Other Study IDs: ITFPEDENDO1
Record Dates: First submitted 2024-07-09; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Growth Alteration; Obesity
Keywords: height; obesity; growth
MeSH Terms: conditions — Obesity | interventions — Body Height; Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- young Turkish males: Aged between 18 - 26 years old Istanbul University students Gender: Male
  Interventions: Other: height and weight measurement
- young Turkish females: Aged between 18 - 26 years old Istanbul University students Gender: Female
  Interventions: Other: height and weight measurement

INTERVENTIONS:
Other: height and weight measurement — Height and weight measurements and socioeconomic status survey
  Other Names: filling out the socioeconomic status survey

SUMMARY:
Current Turkish growth reference charts based on anthropometric measurements of individuals with high socioeconomic status in Istanbul in 1989-2002 (TK2002) had shown an increase of mean adult height (1.4 and 2.7 cm in males and females) compared with 1978. Given recent improvements in nutrition, hygiene and access to preventive health services, it is hypothesized that this positive secular trend may continue. A prior power analysis (95% power) showed that at least 122 subjects of each sex were needed to detect a 1.8 cm height increase (p=0.05) vs TK2002. In 2023-2024 a sample of Turkish young adults (18-26 years) was randomly selected from 65,000 students at Istanbul University, originating from every region of Turkey (TK2024). Height, weight, and socioeconomic status (SES, categorized into four groups) were recorded and body mass index (BMI) was calculated. Adult height and BMI were compared with TK2002 and with young adults of Turkish origin living in the Netherlands measured in 2009 (NL2009).

DETAILED DESCRIPTION:
Study setting A sample of students was randomly selected from 65,000 students at Istanbul University, originating from every region of Turkey in 2023-2024 (TK2024). The inclusion criteria for the study were: (I) age between 18 and 26 years, (II) being a student at Istanbul University, and (III) volunteering to participate in the study. The exclusion criteria were: (I) diagnosis of a chronic disease, (II) a history of surgery that can affect linear growth, (III) diagnosis of growth retardation, (IV) a history of growth hormone administration, (V) having a parent born outside of Turkey, (VI) birth height or weight less than -2 SDS, and (VII) current height or BMI less than -3 SDS or greater than +3 SDS. This study was approved by the Local Ethical Committee of Istanbul Faculty of Medicine and funded by the Scientific Research Projects Coordination Unit of Istanbul University. Voluntary, informed, written consent was obtained from all the participants. The students' medical history, birthplace, high school graduation province, parental education level and occupation and household income were recorded through a questionnaire.

Measurements Standing height was measured with bare feet using a portable stadiometer and documented to the nearest 0.1 cm. Weight was determined in light clothing using a digital scale and recorded to the closest 0.1 kg. Two trained technicians performed all measurements. Height measurements were repeated twice, and the mean value was calculated. If the difference exceeded 0.3 cm, a third measurement was taken, and the average of the two closest values was used. Body mass index (BMI) was calculated as weight (kg) divided by height (m) square .

Classification of socioeconomic status After collecting all the data, the participants were classified into four groups according to socioeconomic status (SES): SES-1 to 4. SES was determined based on the criteria used in previous national growth studies, which were modified to better align with current conditions. This classification is determined by the educational level of both parents and the father's occupation. Meeting all three criteria was necessary for inclusion in the upper levels of the SES. If any of these criteria are not met, individuals were assigned to a lower SES level.

In the present study, the SES assessment questionnaire is derived from the TK2002 questionnaire, with a single modification: the educational level of parents has been increased by one level. This update is based on data from the Turkish Statistical Institute, which reported a 26% average increase in the duration of education in Turkey between 2008 and 2022.

Comparative Analyses To demonstrate the secular trend, a comparison was made between the data from the present study and the data from the 18-year-old age group in the TK2002 study, which served as the basis for the current national growth curves. The data for 18-year-olds in TK2002 were collected from measurements of senior high school students in six affluent districts of Istanbul. In line with the methodology of the present study, TK2002 also categorized participants into four SES groups based on an SES questionnaire.

The technical specifications and measurement methods of the instruments used in this study are identical to those used in TK2002, ensuring comparability and consistency across both studies.

Adult height and BMI were also compared with TK2002 and with young adults of Turkish origin living in the Netherlands measured in 2009 (NL2009). Age, SES, and geographical region were used to conduct subgroup analyses. Age groups were divided into 18-22 and 23-26 years. Separate subgroups were formed for the seven regions of Turkey based on birthplace or high school graduation.

ELIGIBILITY:
Inclusion Criteria:

Age:

Participants must be between 18 and 26 years old.

Student Status:

Participants must be current students at Istanbul University.

Voluntary Participation:

Participants must voluntarily agree to participate in the study and provide informed, written consent.

Exclusion Criteria:

Chronic Disease:

Participants with a diagnosis of any chronic disease are excluded.

History of Surgery Affecting Growth:

Participants with a history of any surgery that could affect linear growth are excluded.

Growth Retardation:

Participants with a diagnosis of growth retardation are excluded.

Growth Hormone Administration:

Participants who have received growth hormone treatment are excluded.

Parental Origin:

Participants with a parent born outside of Turkey are excluded.

Birth Height or Weight:

Participants with a birth height or weight less than -2 standard deviations (SDS) are excluded.

Current Height or BMI:

Participants with a current height or BMI less than -3 SDS or greater than +3 SDS are excluded.

Ages: 18 Years to 26 Years | Sex: All
Age Groups: Adult
Study Population: The study population consists of young adults aged 18 to 26 years who are current students at Istanbul University, representing a diverse demographic background from various regions of Turkey. A total of 465 participants were included in the study, with 217 females and 248 males. The participants were randomly selected from a pool of 65,000 students, ensuring a representative sample of the university's diverse student body. This selection process aimed to capture a wide range of socioeconomic statuses and geographical origins, reflective of the overall Turkish population.
Sampling Method: Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Mean Adult Height (cm) | 01.09.2023- 01.05.2024
  Mean height difference in centimeters between the cohorts (Objective: To compare the mean adult height of young Turkish adults in 2023-2024 (TK2024) with those in 2002 (TK2002) and young adults of Turkish origin living in the Netherlands in 2009 (NL2009))
Change in Body Mass Index (BMI, kg/m²) | 01.09.2023- 01.05.2024
  Mean BMI difference and percentage of participants classified as overweight or obese between the cohorts (Objective: To compare the BMI of young Turkish adults in 2023-2024 (TK2024) with those in 2002 (TK2002) and young adults of Turkish origin living in the Netherlands in 2009 (NL2009)) (BMI was calculated as weight (kg) divided by height (m²), with weight measured using a digital scale (SECA 813, Hamburg, Germany).)

SECONDARY OUTCOMES:
Association between Height and Socioeconomic Status (SES) | 01.05.2024-01.07.2024
  Comparison of mean height across different SES groups
Association between BMI and Socioeconomic Status (SES) | 01.05.2024-01.07.2024
  Comparison of mean BMI across different SES groups
Regional Differences in Height | 01.05.2024- 01.07.2024
  Mean height differences across regions
Regional Differences in BMI | 01.05.2024 - 01.07.2024
  Mean BMI differences across regions ()

CONTACTS AND LOCATIONS:
Overall Officials: Asli Derya Kardelen Al, MD, Study Chair — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)